CLINICAL TRIAL: NCT00403312
Title: Increasing Physical Activity to Aid Smoking Cessation
Brief Title: Increasing Physical Activity as Part of a Smoking Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 381; R01HL068569 (NIH)
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Smoking Cessation
Keywords: Physical Activity; Wellness Programs; Pharmacological Smoking Cessation
MeSH Terms: conditions — Smoking Cessation; Motor Activity | interventions — Tobacco Use Cessation Devices; Exercise

INTERVENTIONS:
Behavioral: Smoking Cessation Behavioral Program
Drug: Nicotine Patch
Behavioral: Physical Activity

SUMMARY:
Cigarette smoking is the most common risk factor for lung cancer, and it increases the risk of developing other cancers, chronic lung disease, and heart disease. A smoking cessation program that incorporates physical activity may be beneficial in improving long-term smoking cessation rates. This study will evaluate the effectiveness of a community-based physical activity program, in combination with nicotine replacement therapy and a behavioral smoking cessation program, at improving cessation rates among sedentary smokers.

DETAILED DESCRIPTION:
Tobacco use is the single most preventable cause of death in the United States, with cigarette smoking accounting for nearly one-third of all cancer deaths each year. While a number of inexpensive and effective smoking cessation methods exist, including the nicotine patch and nicotine gum, smoking rates have not declined in the past few years. Individuals who engage in regular exercise, in addition to participating in a smoking cessation program, are often successful at quitting smoking and reducing post-cessation weight gain. However, past studies on this topic have consisted of highly structured, supervised physical activity, which made study recruitment and long-term adherence difficult. Additionally, these studies generally have had low long-term quit rates, which may be attributed to the lack of a nicotine replacement component. The purpose of this study is to evaluate the effectiveness of a community-based physical activity intervention, in combination with a behavioral smoking cessation program and nicotine replacement, at increasing smoking cessation rates among sedentary adult smokers.

This 7-week study will enroll sedentary or minimally active cigarette smokers. All participants will take part in a behavioral smoking cessation program and will wear a nicotine patch. In addition, they will be randomly assigned to take part in either a community-based physical activity intervention or a wellness control group intervention. All participants will attend sixteen 60- to 90-minute face-to-face counseling sessions and twelve 20-minute telephone counseling sessions. They will also receive twelve informational mailings. Participants in the physical activity intervention will focus on increasing physical activity; the general wellness control group will receive information on general health topics. Outcome measures, including smoking status, physical activity levels, and body mass index, will be assessed at the end of the intervention and at 6- and 12-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Smokes five or more cigarettes each day in the year prior to study entry
* Sedentary or minimally active physical activity level
* Willing to be randomly assigned to either intervention group
* Willing to use the nicotine patch

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant in the year following study entry
* Planning to move out of the area in the year following study entry
* Blood pressure greater than 160/95 mm Hg
* Body weight greater than 140% of ideal body weight
* History of heart attack, stroke, unstable angina, coronary artery bypass grafting, angioplasty, or stent in the 6 months prior to study entry
* Symptomatic peripheral artery disease
* History of congestive heart failure (New York Heart Association [NYHA] Class III or IV)
* Electrocardiogram (EKG) evidence of 2nd or 3rd degree atrioventricular (AV) block
* History of a serious illness that might limit longevity (e.g., significant kidney disease, liver disease, cancer)
* Current substance abuse
* Current alcohol use of more than 21 drinks per week
* Uncontrolled arrhythmia or hyperthyroidism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2003-01

PRIMARY OUTCOMES:
Smoking status (measured immediately post-intervention and at 6- and 12-month follow-up visits)

SECONDARY OUTCOMES:
Changes in self-reported and objective physical activity
Body mass index
Percentage of body fat
Waist circumference (all measured immediately post-intervention and at 6- and 12-month follow-up visits)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D. Ward, PhD, Principal Investigator — University of Memphis
Locations (2):
- United States (2):
  - University of Memphis Center for Community Health, Memphis, Tennessee
  - Department of Preventive Medicine, University of Tennessee Health Science Center, Memphis, Tennessee

REFERENCES:
- [Derived] Stockton MB, Ward KD, McClanahan BS, Vander Weg MW, Coday M, Wilson N, Relyea G, Read MC, Connelly S, Johnson KC. The Efficacy of Individualized, Community-Based Physical Activity to Aid Smoking Cessation: A Randomized Controlled Trial. J Smok Cessat. 2023 May 26;2023:5535832. doi: 10.1155/2023/5535832. eCollection 2023. PMID 37273658